CLINICAL TRIAL: NCT05010265
Title: An Ethical Approach to Detecting Covert Consciousness: Data-Driven Neuroethics for Consciousness Detection (DECODE)
Brief Title: An Ethical Approach to Detecting Covert Consciousness
Acronym: DECODE
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J. Young, M.D., M.Phil, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2021p001738; 1F32MH123001-01 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-08-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Disorder of Consciousness
Keywords: Disorders of consciousness, Advanced neuroimaging
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Use of advanced neurotechnologies to detect consciousness and predict recovery: Treating clinicians, family members (caregivers) and patients recovering from a diagnosis of coma, vegetative state, or minimally conscious state minus (i.e. minimally conscious state without language function)
  Interventions: Other: Clinician Questionnaire; Other: Semi Structured Interviews

INTERVENTIONS:
Other: Clinician Questionnaire — Surveys will serve to identify preferences, expectations and concerns among clinicians and researchers surrounding data-sharing of uncertain diagnostic data generated through investigative neurotechnologies which will then be systematically evaluated.
Other: Semi Structured Interviews — Semi-structured interviews will further serve to identify preferences, expectations and concerns among patients, surrogates, clinicians and researchers surrounding data-sharing of uncertain diagnostic data generated through these investigative neurotechnologies which will then be systematically evaluated.

SUMMARY:
This study aims to develop an ethical approach to developing and deploying novel neurotechnologies to aid in the detection of consciousness and prediction of recovery after brain injury.

DETAILED DESCRIPTION:
Previous studies of patients with disorders of consciousness (DoC) have suggested that conscious patients may be misdiagnosed as unconscious up to 40% of the time when traditional qualitative bedside examination is used (Schnakers et al. 2009, Van Erp et al. 2015, Fins and Bernat 2018). Given the well-established prognostic relevance of early behavioral recovery of consciousness for long-term functional outcomes (Giacino and Kalmar 1997, Giacino 2004, Portaccio et al. 2018, Faugeras et al. 2018, Pincherle et al. 2019), whether or not a patient is considered to be conscious is often the primary determinant of whether life-sustaining therapy is continued and neurorehabilitation is offered. Recent advances in neuroimaging and electrophysiologic neurotechnologies, including functional magnetic resonance imaging (fMRI) and electroencephalography (EEG), have yielded novel methods to aid in detecting and predicting emergence of consciousness in patients with brain injuries. Despite these unprecedented research advances, little is known about ethical concerns surrounding these novel neurotechnologies, about the phenomenological, ontological and ethical valence of conscious states of being without behaving revealed through their lens, or about the attitudes of clinicians, researchers, patients and caregivers regarding their responsible implementation. This study aims to fill these crucial knowledge gaps and to support the development of an evidence-based strategy for ensuring responsible research and translation of novel neurotechnologies to aid in the detection of consciousness and prediction of recovery after brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prior or ongoing participation as subject in a research study using neurotechnologies for diagnosis and prognosis of disorders of consciousness (DoC) at Mass General Brigham
* Patients capable of understanding and answering questions in English
* Patients cble to provide informed consent
* Patients for whom MRI / EEG are administered for clinical detection of consciousness and/or neuroprognostication
* Family member or surrogate caregiver of patients who previously participated or are currently participating in a research study using neurotechnologies for diagnosis and prognosis of DoC at Mass General Brigham.
* Family Members / Surrogates capable of understanding and answering questions in English
* Family Members / Surrogates able to provide informed consent
* Family member or surrogate caregiver of patients for whom MRI / EEG are administered for clinical detection of consciousness and/or neuroprognostication
* Research Investigators involved with research responsibilities in designing or testing neurotechnologies on patients with DoC.
* Clinicians with clinical responsibilities caring for patients in behaviorally unresponsive state, defined as coma, vegetative state (VS), and low-level minimally conscious state (MCS).
* Selected leaders and advisors (Community and Thought Leaders) from brain injury associations and advocacy organizations, and policy-makers involved in decision-making impacting patients with DoC.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disorders of consciousness (DoC)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Surveys and semi-structured interviews | through study completion, an average of 1 year
  Capture and evaluate salient perspectives, preferences and values surrounding the use of advanced neurotechnologies to detect consciousness and predict recovery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Young, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No